CLINICAL TRIAL: NCT02232685
Title: Whole Body Bone Scan vs 18F-Choline PET/CT, Better Detection of Bone Metastases in Prostate Cancer Patients, PROSTAGE I
Brief Title: Whole Body Bone Scan vs 18F-Choline PET/CT in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mike Allan Mortensen, MD, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAM_PROSTAGE1
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Staging; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Choline PET/CT (Experimental): 18F-Choline PET/CT
  Interventions: Device: 18F-Choline PET/CT

INTERVENTIONS:
Device: 18F-Choline PET/CT — 18F-Choline PET/CT

SUMMARY:
Prostate cancer is currently the leading newly diagnosed cancer in the industrialized world. Treatment of prostate cancer is highly dependent on the stage of the disease. Current methods for staging are known to be inaccurate. Prior studies from our department suggest that PET/CT is useful in staging of bone metastases in patients with prostate cancer. The aim of this study is to test the usefulness of Choline PET/CT for the staging of bone metastases compared to current standard methods in patients with newly diagnosed prostate cancer.

Better initial staging will result in better treatment of the individual patient. If we are able to develop a more accurate method of staging patients with undetected metastases on current staging will be spared of the side-effects associated with current treatment - impotence, incontinence, radiation damage etc.

DETAILED DESCRIPTION:
1. Introduction. Cancer of the prostate (PCa) is currently the leading newly diagnosed cancer and the second most common cause of cancer deaths among men in the industrialized world . In Denmark alone more than 4000 men are yearly diagnosed with PCa . As PCa primarily affects elderly patients, one can assume that PCa will become one of the most important medical issues in the developed world due to the already high incidence combined with a growing population of elderly men.

   The aetiology of the disease is not well understood. In its most common form PCa evolves from the glandular tissue of the prostate. Metastatic spread will most commonly happen as lymphogenous spread to the regional lymph nodes or as haematogenous spread to the red bone marrow .

   Intended curative treatment of PCa is associated with considerable side effects, in particular incontinence, impotence and radiation damage to the surrounding tissues. Furthermore, over 30% of patients with organ-confined disease, which was treated with radical prostatectomy, will have biochemical relapse within 10 years . Relapse may be due to local recurrent disease suggesting poor surgical quality or poor initial staging with undetected metastases at the time of treatment.

   At diagnosis patients are stratified as having low, intermediary or high risk of dissieminatio according to D'Amico. Patients with intermediate or high risk of dissemination will be examined further with whole-body bone scintigraphy (WBS) and pelvic lymph node dissection (PLND).
2. Background. 2.1. Current staging and limitations. WBS has been the examination of choice for evaluation of potential dissemination to bone. WBS utilizes 99mTc-labeled methylene diphosphonate (99mTc-MDP) that binds to the bone matrix formed by the osteoblasts. Gamma cameras detect the γ-radiation emitted by the decaying tracer thereby creating a 2-dimentional image depicting local osteoblast activity .

   Several limitations apply to the use of WBS in staging of patients with PCa. Sensitivity has reported as low as 39% in lesion-based analysis in patients with a low number of lesions . This combines with a low sensitivity due to many equivocal lesions caused by other bone pathology than metastasis.

   Sensitivity and specificity is improved by the use of single-photon emission computed tomography (SPECT), where the same tracer as with WBS is used to generate a three-dimensional image using a rotating gamma camera. This method also gives better anatomical information on the exact position of a potential metastasis.

   The examination of choice for the evaluation of potential metastases to lymph nodes is extended PLND . This procedure is done either prior to radiotherapy or during prostatectomy in patients with intermediate or high risk of dissemination. The optimal extent of the dissection is debated. The extended PLND performed at our institution includes the nodes in the obturator fossa, the nodes over the external iliac artery and vein, the nodes around the internal iliac artery and the nodes along the common iliac artery up to the crossing of the ureter. This dissection is assumed to include approximately 75% of lymph nodes known to harbor primary prostatic lymph node metastases . Extended PLND is surgically demanding with risk of lymphocele formation, infectious complications and severe bleeding due the lymph nodes' close proximity to the large vessels in the pelvis. All in all extended PLND is perhaps the best option for lymph node staging of PCa but it cannot be considered as optimal due to the above-mentioned issues.

   2.2 Positron Emission Tomography (PET). Positron Emission Tomography combined with Computerized Tomography (PET/CT) is a well-established tool in diagnosing and staging of several types of cancer . PET is an imaging technique where pairs of gamma rays emitted by positron-emitting radionuclide tracer are detected, producing a three-dimensional image of tracer concentration based on the amount of gamma rays emitted. The radioactive tracer is coupled to a biologically active molecule depending on the organ or metabolic process of interest . These images can then be fused with CT to create a combined functional and high-resolution anatomical image. Several tracers have been developed for use in cancer diagnostics and staging. As of now, PET/CT has no generally accepted role in the diagnosing or staging of PCa neither in Europe nor in the US .

   2.2.1 Choline. Choline is a precursor for phosphatidylcholine, a phospholipid that is integrated in the cell membrane making it a marker for cell membrane turnover and metabolism . 11C-Choline was first used as a PET tracer in 1997 . Since then many studies have been performed with 11C-Choline and later 18F-Choline (FCH) having approximately the same properties as 11C-Choline, but with a longer half-life (110 min vs. 20 min) making it more versatile in every-day use. A recent study from our department tested the use of FCH-PET/CT in detecting lymph node metastasis in 210 patients with PCa . The study concluded that FCH-PET/CT was not ideally suited for lymph node staging but could give additional information about bone metastasis. Several other investigators have also implied this , . A likely reason for the better detection of metastasis to the bone is that bone metastasis in an early stage is actually bone-marrow metastases rather than bone matrix metastasis and that it most likely that bone-marrow metastases proceed to bone matrix metastases. These will not be detectable by WBS (and probably not by CT and MRI either). Larger prospective series on the use of FCH-PET/CT for imaging of bone metastasis in PCa-patients have not yet been produced.
3. Trial objective. To compare the diagnostic accuracy in detecting bone metastases of WBS, SPECT and FCH PET/CT in 280 patients with newly diagnosed PCa with intermediate or high risk of disseminated disease
4. Method. The patients will have two scans performed, first one with two acquisitions using only one administration of tracer i.e. a WBS followed by a SPECT acquisition and on another day a FCH-PET/CT. Image acquisition will be performed approximately 60 min after intravenous injection of the tracer.

The scans are performed in random order within three weeks and the images interpreted by a specialist in nuclear medicine and a specialist in radiology. Patients who already have had WBS performed will only have a FCH-PET/CT performed.

Images are interpreted based on visual evaluation with supplementary measurements of Standardized uptake values (SUV).

In case of agreement between the scans, the patient will proceed to clinical treatment as usual. In case of disagreement between the three modalities a MRI will be performed on the lesion of interest. If the results after MRI are still inconclusive a bone biopsy with emphasis on getting marrow tissue as well as bone matrix, will be performed. This will in many cases not be possible due to the size of the lesion and in these cases MRI will serve as reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically verified PCa and
* Written consent and
* PSA ≥ 20 ng/mL and/or
* Gleason score > 6 and/or
* cT-stage ≥ cT2c

Exclusion Criteria:

* Withdrawal of consent or
* Other active malign disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Metastases to bone (yes/no) | 1 day (At the time of scan interpretation)

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospiatal, Odense, Denmark